CLINICAL TRIAL: NCT00639093
Title: A Virtual Arm to Stop Smoking. A Comparative Study
Brief Title: A Virtual Arm to Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Quebec en Outaouais (Other)
Responsible Party: Principal Investigator, Stephane Bouchard, Professor, Universite du Quebec en Outaouais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRAP-CRC-cyberpsychologie
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2009-07-31 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Cigarette Smoking
Keywords: cigarette smoking; psychoeducational and motivational program; virtual reality
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): All participants will receive an eight-session psychoeducational and motivational program. During the first four weeks, all participants will be immersed in virtual reality (VR).
  During the immersions in VR, 45 of the participants will use a virtual reality arm to catch and crush virtual cigarettes (on a computer).
  Interventions: Behavioral: psychoeducational / motivational combined with crushing
- 2 (Active Comparator): All participants will receive an eight-session psychoeducational and motivational program. During the first four weeks, all participants will be immersed in virtual reality (VR).
  During the immersions in VR, the 45 participants in the control condition will use a virtual reality arm to catch and crush virtual fruits (on a computer).
  Interventions: Behavioral: psychoeducational / motivational combined with control

INTERVENTIONS:
Behavioral: psychoeducational / motivational combined with crushing — All participants will receive an eight-session psychoeducational and motivational program. During the first four weeks, all participants will be immersed in virtual reality (VR).
  During the immersions in VR, 45 of the participants will use a virtual reality arm to catch and crush virtual cigarettes (on a computer).
  Arms: 1
Behavioral: psychoeducational / motivational combined with control — All participants will receive an eight-session psychoeducational and motivational program. During the first four weeks, all participants will be immersed in virtual reality (VR).
  During the immersions in VR, the 45 participants in the control condition will use a virtual reality arm to catch and crush virtual fruits (on a computer).
  Arms: 2

SUMMARY:
The investigators reported in a pilot study presented at last year's Cybertherapy Conference (Girard & Turcotte, 2007) that using an action-cue exposure strategy in virtual reality (ACE-VR; crushing virtual cigarettes) might be useful in the treatment of tobacco addiction.

The investigators are pursuing research in this area with a randomized control trial based on 90 smokers who will receive a brief psychosocial smoking cessation program (25 people are enrolled so far and we expect to finish the study before the conference). During the first four weeks of an eight-session psychoeducational and motivational program, all participants will be immersed in VR. During the immersions in VR, 45 of the participants will use a virtual arm to catch and crush virtual cigarettes. The other half of the sample will use the virtual arm to catch virtual fruits (control condition).

The smoking frequency, and abstinence, will be assessed with a daily diary and exhaled carbon monoxide tests (the CO2 tests will provide an objective confirmation of the abstinence reported in the diaries). The success the program will be compared based on the number of subjects who quitted or reduced their smoking frequency. The severity of addiction will be assessed with two questionnaires, the Fagerstrom and the Horn tests. Craving and withdrawal effects will be measured with the Minnesota Nicotine Withdrawal Scale (MNWS) and the Brief Questionnaire of Smoking Urges (QSU-Brief) at the baseline and at the visits from weeks 1 through 4, 6, 12 and at the end of the program. Before the VR immersion, the Immersive Tendencies Questionnaire will be administered and after each VR session participants will fill two questionnaires addressing presence and cybersickness. The comparative impact of both treatments will be tested with repeated measures ANOVAs (and planned contrasts) with sufficient power to detect medium effect sizes.

The main goal of our study is show that crushing virtual cigarettes can boost the impact of a behavioural program dedicated to cigarette addiction.

DETAILED DESCRIPTION:
A detailed description is available, in French, by contacting stephane.bouchard@uqo.ca.

ELIGIBILITY:
Inclusion Criteria:

* adult smoker
* aged 18 - 65
* willing to stop smoking
* at least 10 cigarettes per day in the last year

Exclusion Criteria:

* receiving concomitant treatment for smoking (e.g., patches or varenicline)
* weight problems : Body Mass Index < 15 kg or > 45.5 kg
* suffering from a mental disorder, such as major depression, schizophrenia, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — G.R.A.P.; Stephane Bouchard, Ph.D., Study Chair — U.Q.O.
Locations (1):
- GRAP - Clinique de psychologie au travail, Jonquière, Quebec, Canada

REFERENCES:
- [Background] Girard, B., & Turcotte, V. (2007). A virtual arm to stop smoking, a perceptual learning experiment. In N. Appel & H. Hoffman (Chairs), Addictions. Symposium presented at the Cybertherapy 12 Conference, in June in Washington, D.C.
- [Background] Martin RA, Rohsenow DJ, MacKinnon SV, Abrams DB, Monti PM. Correlates of motivation to quit smoking among alcohol dependent patients in residential treatment. Drug Alcohol Depend. 2006 Jun 9;83(1):73-8. doi: 10.1016/j.drugalcdep.2005.10.013. Epub 2005 Nov 28. PMID 16314049
- [Derived] Girard B, Turcotte V, Bouchard S, Girard B. Crushing virtual cigarettes reduces tobacco addiction and treatment discontinuation. Cyberpsychol Behav. 2009 Oct;12(5):477-83. doi: 10.1089/cpb.2009.0118. PMID 19817561
- See also: Click here for more information about this study about the virtual arm — http://www.grap.ca/
- See also: Click here for more information about clinical applications of virtual reality — http://w3.uqo.ca/cyberpsy
- See also: For more information about using VR to treat smoking — http://www.virtuallybetter.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical clinic in the province of Quebec.
Groups:
- VR - Cigarettes: All participants will receive an eight-session psychoeducational and motivational program. During the first four weeks, all participants will be immersed in virtual reality (VR).
  During the immersions in VR, 45 of the participants will use a virtual reality arm to catch and crush virtual cigarettes (on a computer).
- VR - Balls (Control): All participants will receive an eight-session psychoeducational and motivational program. During the first four weeks, all participants will be immersed in virtual reality (VR).
  During the immersions in VR, the 45 participants in the control condition will use a virtual reality arm to catch and crush virtual fruits (on a computer).
Period: Overall Study
Arm/Group | VR - Cigarettes | VR - Balls (Control)
Started | 45 (45) | 46 (46)
Completed | 45 (45) | 46 (46)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VR - Cigarettes | VR - Balls (Control) | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Categorical [Count of Participants; unit: Participants] — Aged above 18.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 45 | 46 | 91
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Canada | 45 | 46 | 91
Nicotine addiction [Number; unit: Participants] — As stated in the Eligibility Criteria, participants had to be smokers (10 cigarettes per day minimum) wanting but incapable to quit.
  Participants | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Self-report Measure of Abstinence in the Last 7 Days, Averaged Over Four Weeks, and Confirmed by Urine Samples.
Description: Participants completed a daily diary to record the number cigarettes smoked during the day. No cigarette smoked during 7 days = abstinence. To be counted as real abstinence, the participant had to smoke zero cigarettes during four weeks and confirmed by zero nicoting in the unrine sample.
  Six measurement times were used to assess if zero cigarettes has been smoked in the last 4 weeks prior to the study (Week 1), during the first four weeks (Week 4 measurement point) and so on for a blok of four weeks ending at each measurement point (e.g., four weeks before the 12-month follow-up).
Time Frame: Weeks 1, 4, 6, 12, 24 and 12-month follow-up
Measure: Number; unit: participants
Arm/Group | VR - Cigarettes | VR - Balls (Control)
Number analyzed (Participants) | 45 | 46
participants | 45 | 46

2. Secondary Outcome: Tiffany's Urge to Smoke Questionnaire
Time Frame: Weeks 1, 4, 6, 12, 24 and 12-month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | VR - Cigarettes | VR - Balls (Control)
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 0/45 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes